CLINICAL TRIAL: NCT00474162
Title: Observational Pilot Study of the Effect of Intravenous Saline or Pentastarch on Coagulation in Women Having an Elective Cesarean Section
Brief Title: The Clotting Effects of Pentastarch and Normal Saline in Obstetric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Children's & Women's Health Centre of British Columbia (Other)
Responsible Party: Dr. Joanne Douglas, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H06-03374
Record Dates: First submitted 2007-05-14; First posted 2007-05-16 (Estimated); Last update posted 2008-02-21 (Estimated); Status verified 2008-02

CONDITIONS: Elective Cesarean Section
Keywords: Cesarean section; coagulation changes
MeSH Terms: interventions — Hydroxyethyl Starch Derivatives; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Pentaspan® — 15 ml/kg of starch solution, approximately 1 litre
Drug: Normal Saline — 15 ml/kg of either saline solution, approximately 1 litre

SUMMARY:
Pregnant women are more likely to form clots than non-pregnant women as pregnancy increases the clotting factors present in the blood. This helps to prevent excess bleeding (hemorrhage) at the time of delivery. Hemorrhage occurs in 5-15% of pregnancies throughout the world, even when delivery is by cesarean section. When hemorrhage occurs the anesthesiologist will normally administer fluids into the woman's vein (intravenously) rapidly to replace the blood that the woman has lost. Two types of fluids are commonly used. One is a salt water solution (saline) and the other is a starch water solution (pentastarch). Use of either or both of these solutions is common during hemorrhage.

These same solutions (salt water solution and starch solution) are used at BC Women's Hospital during spinal anesthesia to prevent and treat low blood pressure (a common side effect of spinal anesthesia). This is standard practice whether you are in this study or not. You may also be given, depending on the anesthesiologist's preference, a drug (vasopressor) that causes the blood vessels to become narrow (constrict) to prevent or treat the low blood pressure. Whether you agree to be part of the study or not, your anesthesiologist will be watching your blood pressure closely throughout your operation and if your blood pressure becomes low he/she will treat it as is normally done.

Low blood pressure will also occur during hemorrhage. It is therefore important that we determine whether the starch solution, which is more effective than the salt solution in preventing low blood pressure during spinal anesthesia, does or does not affect clotting.

Research in non-pregnant adults (male and female) has found that laboratory tests of blood clotting change with these solutions. For saline the evidence in some studies suggests that the blood may clot better than normal while other studies suggest the opposite (does not clot as well). In pregnant and non-pregnant adults the blood does not clot as well with certain starch solutions. The starch solution used at BC Women's Hospital is called pentastarch and no research has looked at its effect on clotting in pregnant women. In non-pregnant adults pentastarch has less effect on clotting than other starch solutions.

The purpose of the study is to see how pentastarch (starch solution) and normal saline (water with salt in it) given at the time of spinal anesthesia for elective cesarean section affect the ability of pregnant woman's blood to clot.

DETAILED DESCRIPTION:
Study patients will be randomized to one of two groups. One group will receive saline solution (salt water) and the other group will receive the pentastarch solution. Neither the patient, the anesthesiologist, the obstetrician nor nurses will know which group the patient is in.

All women who participate in the study will have an intravenous. Once the tube is in the vein, a blood sample will be taken from it before an intravenous solution is started. The amount of blood taken will be approximately 1 tablespoon (15mL). This is not part of routine care but is part of the study. This blood will be checked to see how well it forms a clot. The study solution (15 ml/kg of either saline or starch solution, approximately 1 litre) will then be attached to the intravenous. Once the patient is in the operating room and the spinal anesthetic has been given the remainder of the study solution will be given very rapidly over 10 minutes into the vein. Once the study solution has been given, the patient will receive a saline solution through their intravenous at a rate determined by the anesthesiologist according to their normal practice.

Five minutes after the study solution is given, a further blood sample (15 mL) will be taken from the intravenous and it will be tested the same as for the first blood sample. A third blood sample will be taken approximately 85 minutes later. As these blood samples will be taken from the intravenous, the patient will not have to have a needle inserted to take them. Approximately 10% of the time it may not be possible to take the blood sample from the intravenous. If this should happen the investigator or the anesthesiologist will want to take the blood sample from the opposite arm to the intravenous. The patient will be told that this is going to happen and can withdraw from the study at that time. This will not affect any further care that the patient receives. To minimize discomfort if blood is taken from the opposite arm the skin will be made numb with local anesthetic.

You will be treated the same as any woman having a cesarean section under spinal anesthesia with the exception that

1. the patient and the anesthesiologist will not know which study solution is being given and 2 three blood samples will be taken - to total 3 tablespoons (total: 3x1 tablespoon).

For the purposes of the study we will be using the information collected about the patient in the normal course of the anesthetic, including the total amount of fluid that received during cesarean section, the need for, type and amount of any medication during the cesarean section, and an estimate of the total amount of blood lost during the operation. These are in addition to the results of the laboratory tests of clotting.

There is no extra time or cost involved for the patient.

ELIGIBILITY:
Inclusion Criteria:

* aged 19 years or over
* having an elective cesarean section under spinal anesthesia
* at least 36 weeks gestation
* in general good health

Exclusion Criteria:

* blood does not clot normally
* taking heparin or Aspirin® (acetylsalicylic acid) within 7 days of surgery
* high blood pressure
* expecting twins
* any heart abnormality (including heart failure)
* kidney or liver disease
* known allergy to hydroxyethylstarch, corn, starch or any drugs
* insulin dependent diabetes
* aged less than 19 years
* do not understand English
* having emergency surgery

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2007-05; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
TEG (clotting) parameters at baseline, 5 minutes & 90 minutes post-infusion | During surgery

SECONDARY OUTCOMES:
Changes in INR, APTT and estimated blood loss | During surgery

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Douglas, MD, Principal Investigator — University of British Columbia; Jason Ford, MD, Study Director — University of British Columbia; Roanne Preston, MD, Study Director — University of British Columbia; Rhona Siegmeth, MBChB, BSc, FRCA, Study Director — University of British Columbia
Locations (1):
- BC Women's Hospital, Vancouver, British Columbia, Canada